CLINICAL TRIAL: NCT04787315
Title: Reaching Clinical Recommendations for Intensity of Post-stroke Rehabilitation Using an Activity Circuit Implemented With a Change Agent
Brief Title: Reaching Clinical Recommendations for Intensity of Post-stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Cyril Duclos, Researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRIR-1423-0719
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive rehabilitation without workstation (Active Comparator)
  Interventions: Behavioral: Conventional intensive functional rehabilitation
- Intensive rehabilitation with workstations (Experimental)
  Interventions: Device: Conventional intensive functional rehabilitation + Workstations

INTERVENTIONS:
Device: Conventional intensive functional rehabilitation + Workstations — Equipment will be provided to participants where they can do exercises to increase their motor abilities at the lower limbs, trunk and upper limbs, in addition to conventional intensive functional rehabilitation
  Arms: Intensive rehabilitation with workstations
Behavioral: Conventional intensive functional rehabilitation — Includes rehabilitation interventions provided by professionnals (OT, PT, speech language therapy, neuropsychologists...)
  Arms: Intensive rehabilitation without workstation

SUMMARY:
The project aims to implement workstations for mobility training during intensive inpatient rehabilitation to increase the level of motor activity of individuals with hemiparesis due to stroke

ELIGIBILITY:
Inclusion Criteria:

* Receving intensive rehabilitation care for hemiparesis due to stroke in our rehabilitation facility (IRGLM)

Exclusion Criteria:

* Cognitive deficits preventing participation to rehabilitation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-05 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Actimetry | In the third or fourth week of rehabilitation
  Measure of acceleration data of the paretic lower and upper-limbs by means of an accelerometer (actigraph (r)) placed at the ankle and wrist during seven consecutive days

SECONDARY OUTCOMES:
Gait speed | Baseline, pre-intensive rehabilitation
  Measured using the 10-meter walking speed test
Balance capacities | Baseline, pre-intensive rehabilitation
  Measured using the MiniBESTest or Berg Balance scale according to abilities
Gross manual dexterity | Baseline, pre-intensive rehabilitation
  Measured using the Box and Block test
Gait speed | End-measure, at the end of rehabilitation
  Measured using the 10-meter walking speed test
Balance capacities | End-measure, at the end of rehabilitation
  Measured using the MiniBESTest or Berg Balance scale according to abilities
Gross manual dexterity | End-measure, at the end of rehabilitation
  Measured using the Box and Block test

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Duclos, PhD, Principal Investigator — CIUSSS Centre-Sud-de-l'ile-de-Montréal
Locations (1):
- CIUSSS centre-sud-de-l'ile-de-Montréal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No